CLINICAL TRIAL: NCT06046859
Title: Can Immediate Post-injury Fluoxetine Improve the Recovery Trajectories of Victims in Bodily Trauma?
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB202301506
Record Dates: First submitted 2023-09-05; First posted 2023-09-21 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Musculoskeletal Injury
MeSH Terms: interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Researchers collecting survey data will be blinded to patients' intervention status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Subjects randomized to get Fluoxetine therapy (Experimental): Subjects will be randomized to take Fluoxetine (10mg by mouth per day for first 14 days then 20 mg by mouth for 9 months). The randomized drug will be prescribed by the study team on the day of randomization so that the patient may be monitored for side effects during the remainder of their hospitalization. The patient will be prescribed the randomized medication on the day of discharge and a 90 day supply will be provided by the inpatient research pharmacy at the 2 week, 3 month, and 6 month follow-up visits
  Interventions: Drug: Fluoxetine
- Subjects randomized to Placebo (Active Comparator): When a patient is enrolled, the inpatient research pharmacy will dispense the appropriately randomized medication in a visually similar, over-encapsulated form as Fluoxetine
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluoxetine — Subjects will be randomized to take Fluoxetine (10mg by mouth per day for first 14 days then 20 mg by mouth for 9 months). The randomized drug will be prescribed by the study team on the day of randomization so that the patient may be monitored for side effects during the remainder of their hospitalization. The patient will be prescribed the randomized medication on the day of discharge and a 90 day supply will be provided by the inpatient research pharmacy at the 2 week, 3 month, and 6 month follow-up visits
  Arms: Subjects randomized to get Fluoxetine therapy
Drug: Placebo — When a patient is enrolled, the inpatient research pharmacy will dispense the appropriately randomized medication in a visually similar, over-encapsulated form as Fluoxetine
  Arms: Subjects randomized to Placebo

SUMMARY:
With this prospective double-blinded, placebo controlled clinical trial we hypothesize that immediate (post-injury) intervention with Fluoxetine will prevent/mitigate the development of negative psychiatric symptomology such as PTSD and depression for victims of bodily trauma. We also hypothesize that immediate use of Fluoxetine will decrease subjects' pain, pain interference and opioid use without changing our standard of care post-injury pain medication regimen. Enrolled subjects will be randomized to Fluoxetine or placebo at their index hospitalization.

DETAILED DESCRIPTION:
Upwards of 40-85% survivors of bodily trauma (in the civilian world most commonly motor vehicle accidents, falls and assaults), develop moderate to severe negative psychiatric symptomology following their injuries. (2,7) This symptomology can persist for years; at least 20% of patients with musculoskeletal trauma, specifically, display symptomology consistent with post-traumatic stress disorder (PTSD) symptomology up to three years following their injury. (8) Poor mental health outcomes are an independent risk factor for poor physical and social outcomes. (9,10) These symptoms, which are highly impairing, are complicated and heightened by loss of work/income following trauma, limited financial and social resources, and a large percentage of the population being uninsured/underinsured. Research has demonstrated that the pressures of poverty and low socioeconomic status alone predispose to PTSD symptomology and poor coping mechanisms, and this is compounded by decreased ability to obtain and pay for mental health care by those impoverished. There are significant barriers to mental health care for many adults, and these hurdles are even more insurmountable for those under or uninsured, minorities, and those in rural communities. (11) Very few victims of trauma who screen positive for psychological disorder receive mental health services following injury (12% at 3-months from injury), and if so, it is far removed from the injury (22% at 24-months from injury).

ELIGIBILITY:
Inclusion Criteria:

* Admitted to UF Health for trauma resulting in:

  * One or more extremity fractures requiring surgery
  * Pelvic Fracture
  * Chest/abdominal Injury requiring intervention in operating room
* Polytrauma (multiple organ systems/multiple fractures) or Beck Depression Inventory (BDI-II) ≥ 14

Exclusion Criteria:

* Severe Traumatic Brain Injury or cognitively not able to participate in surveys. (Glasgow Coma Scale 3-8)
* Other psychiatric conditions on current medical management (SSRI)
* Incarceration or Pregnancy
* Expected Injury Survival of less than 90 days
* Medical or physical condition in opinion of investigators that would preclude safe study participation
* Unable to provide informed consent due to language or other barriers
* Current or previous substance abuse (excluding cannabinoids and alcohol)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Beck Dression Inventory survey, in the post injury period for patients with musculoskeletal trauma. | Baseline up to 12 months
  BDI-II Beck Depression Inventory: higher score means worse outcome; 0-63.

SECONDARY OUTCOMES:
Patient reported pain scores, PROMIS Pain Interference, will be recorded at each visit. | Baseline up to 12 months
  PROMIS PI: Pain Interference; A score of 50 is average; Adaptive so no minimum/maximum values.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Hagan, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided